CLINICAL TRIAL: NCT02030197
Title: Effects of an Educational Socialization Program Designed to Improve Self-Efficacy and Subsequent Effects on Decreasing Loneliness and Depression Among People With Multiple Sclerosis
Brief Title: Impact of CRISP on Self-Efficacy, Loneliness, and Depression
Acronym: CRISP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Principal Investigator, J. Tamar Kalina, Program Manager, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S14-00572
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRISP program (Active Comparator): educational and socialization program
  Interventions: Behavioral: CRISP Program
- Control Group (Placebo Comparator): no treatment control group
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: CRISP Program — Educational program to improve self-efficacy, loneliness and depression
  Arms: CRISP program
Other: Control Group — no treatment
  Arms: Control Group

SUMMARY:
The purpose of this study is to examine the effects of an innovative program, entitled CRISP (Community Integration for Socially Isolated Patients), on improving self-efficacy and assessing whether improved self-efficacy helps to reduce depression and loneliness of people with MS.

DETAILED DESCRIPTION:
Whether CRISP increases self-efficacy while decreasing loneliness and depression

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years old.
* Must have a definitive diagnosis of MS by a physician.
* Must understand English at 6th grade level since the CRISP program requires participants to comprehend the educational information presented in English.
* Agree to participate in 12 group sessions over 12 weeks;
* Must have the ability to complete questionnaires in English since the outcome measures used for the study are in English.
* Must be able to commute to the site destinations

Exclusion Criteria:

* Have an actively psychotic Axis I disorder.
* Have a significant Axis II disorder of borderline personality disorder or schizoid personality disorder.
* Have a diagnosis of another neurological condition aside from MS.
* Inability to comply with study requirements/visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Multiple Sclerosis Self-Efficacy Scale (MSSS) | Change from Baseline to week 12
  The Multiple Sclerosis Self-Efficacy Scale (MSSS) is designed to measure self-efficacy in people diagnosed with MS. The MSSS incorporates aspects of social interaction and themes related to beliefs of control over future events, which is based on Bandura's definition of self-efficacy (Rigby et al., 2003). The MSSS is a 14 item, six-point Likert scale and participants are asked to rate their level of agreement or disagreement for each item on the scale ranging from 'strongly disagree' (1) to 'strongly agree' (6). Examples of questions include "sometimes I feel embarrassed in public places" or "I have as much independence as I need." Scores can range from 14 (low self-efficacy) to 84 (high self-efficacy).

SECONDARY OUTCOMES:
UCLA Revised Loneliness Scale | Change from Baseline to week 12
  The UCLA Revised Loneliness Scale was developed to assess subjective feelings of loneliness and is widely used in loneliness research. The scale consists of 20 questions about loneliness asking participants to rate each question from 1 (never) to 4 (always), higher scores indicating greater degrees of loneliness.
Chicago Multiscale Depression Inventory (CMDI) | Change from Baseline to week 12
  The Chicago Multiscale Depression Inventory will be used to assess symptoms of depression. The CMDI is a 50-item self-report measure that includes three subscales representing different types of depression symptoms: vegetative, mood, and evaluative. Each item on the scale consists of a single word or brief phrase describing feelings or experiences and participants rate each item on a Likert scale from 1 (not at all) to 5 (extremely).
Performance Scales (PS) | Change from Baseline to week 12
  The Performance Scales (PS) is a self-reported measure of MS disease status assessing mobility, hand function, vision, fatigue, cognitive symptoms, bladder/bowel, sensory symptoms, spasticity, pain, depression, and tremor/coordination. Each scale of the PS (with the exception of the mobility scale) is a 6 item ordinal scale and participants are asked to describe their functioning in each area as compared to before they developed MS. Scores range from normal (0) to total disability in specified area (5) with higher scores indicating greater perceived disability. The mobility scale has a range from normal (0) to total gait disability or bedridden (6) and asks participants to choose the category that describes their walking ability in the past four weeks.
Community Integration Questionnaire (CIQ) | Change from Baseline to week 12
  The Community Integration Questionnaire (CIQ) was developed to assess community integration after an injury with questions about home integration, social integration and productive activities. The CIQ is a 15 item self-report measure. The basis for scoring is by the frequency of performing specific activities and providing subtotals for each category of community integration as well as an overall score.

CONTACTS AND LOCATIONS:
Locations (1):
- NYU MS Center, New York, New York, United States